CLINICAL TRIAL: NCT02006082
Title: Readmissions to Hospital and Patient Satisfaction Among Patients With Chronic Obstructive Pulmonary Disease After Telemedicine Video Consultation - a Pilot Project
Brief Title: Readmissions to Hospital Among Patients With COPD After Telemedicine Video Consultation - a Pilot Project
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: SUS-IDPVO2011/50; SUS-IDPVO2011/50COPD (Other: SUS)
Record Dates: First submitted 2013-09-13; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Telemedicine video-consultation (TVC); Re-admission to hospital; Time to re-admission; Length if hospital stay; Patient satisfaction; Chronic obstructive pulmonary disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COPD patients followed after TVC: All COPD patients living in the southern part of Rogaland county in Western Norway, with a habitual value of FEV1 < 50%, who were monitored at home by TVC following discharge after emergency hospitalization for COPD exacerbation at Stavanger University Hospital, or who had tele-monitoring at home under outpatient treatment for acute COPD deterioration during the pilot project period (16th April 2010 - 31st December 2011). The telemedicine equipment consisted of a computer with a web camera with a microphone, through which the patient at home and the specially trained nurse in hospital were able to communicate, and also comprised requisites to measure the patient's oxygen saturation and heart rate, and to perform a spirometry.
  Interventions: Device: Telemedicine video-consultation (TVC)

INTERVENTIONS:
Device: Telemedicine video-consultation (TVC) — All patients enrolled in the study, were previously monitored by TVC, and the number and length of hospital stays within 6 and 12 months following TVC were compared to similar numbers before TVC in comparable time periods. Thus, TVC is actually not to be considered as an intervention.
  Other Names: Video-conferencing in Telemedicine

SUMMARY:
The purpose of this study was to evaluate the effects of telemedicine video-consultation (TVC) on the frequency of hospital re-admissions during 12 months follow-up after TVC among patients with chronic obstructive pulmonary disease (COPD). Our secondary aims were to assess the impact of TVC on the length of recurrent hospital stays and time to re-admission within 12 months follow-up after TVC. We also wanted to evaluate the patient satisfaction related to TVC.

DETAILED DESCRIPTION:
The study is conducted as a retrospective uni-center observation study of a population of COPD patients who after discharge from hospital for acute COPD exacerbation, or during outpatient treatment for acute COPD exacerbation, was monitored for 2 weeks by TVC during a pilot project period from 16 April 2010 to 31 December 2011. To study a possible change in amount of hospital admissions we have compared the frequencies and durations of such events before and after TVC in comparable time periods.

A detailed patient history comprising demographic data, social status, smoking habits, body mass index (BMI), use of medication, co-morbidity and the habitual lung function were registered. Dates of admittance and discharge were noted. Retrospectively, medical records were scrutinized for re-admissions due to COPD exacerbations at 12 months follow-up. Frequency of and date of re-admissions, length of hospital stay, and clinical data were recorded. Also frequency of admission due to COPD exacerbation and length of hospital stay(s) during the last 12 months prior to the TVC were recorded, and date of last discharge was noted. Finally, all patients were encouraged to complete a questionnaire concerning patient satisfaction and impact on patient's quality of life. All answers were registered anonymously.

Data were entered to a database by one trained nurse and monitored by another person, who compared data entered into the registry against predefined rules for range or consistency with other data fields in the registry. All patients who had been monitored by TVC during the pilot project period, gave informed consent to participate in the observational study, and no patient was lost to follow-up.

Continuously distributed variables of baseline characteristics were given as mean + SEM, while variables with more skewed distributions were given as median and upper and lower quartiles.

The Shapiro-Wilk test for normality was performed to study the distribution of parameters. A chi-square test was applied to compare the frequency of re-admissions during 12 months following TVC to the frequency of hospital admissions during the last 12 months prior to TVC. The total number of days in hospital during the last 12 months prior to TVC was compared to number of days in hospital during 12 months following TVC by a paired t-test. Differences in baseline characteristics between patients who were re-admitted and those who were not, were analyzed by a Two-sample Student's T-test, or in case of non-normality, by the Mann-Whitney Rank Sum test.

The number of days to re-admission following TVC as compared to number of days from last discharge to date of index admittance was displayed in a Kaplan Meier plot, with a hazard ratio (HR) calculation by a by a Cox regression analysis.

A statistically significant level of p < 0.05 was applied for all tests. All statistical analyses were performed using the statistical package of SigmaPlot Version 12.

Power calculations have not been performed for the purpose of this pilot study, because of too many unknown factors. The results of this study will form the basis of power calculations for a future prospective randomized study.

ELIGIBILITY:
Inclusion criteria:

* All COPD patients living in the southern part of Rogaland county in Western Norway, with a habitual value of FEV1 < 50%, who were monitored at home by TVC following discharge after emergency hospitalization for COPD exacerbation at Stavanger University Hospital or DMC in Egersund, or who had tele-monitoring at home under outpatient treatment for acute COPD deterioration during the pilot project period
* Written informed consent was obtained

Exclusion critera:

* Previously inclusion in the study
* Unwillingness to participate
* Residence in service housing with care or in nursing homes
* Inability to communicate

Ages: 40 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All COPD patients living in the southern part of Rogaland county in Western Norway, who were monitored at home by TVC following discharge after emergency hospitalization for COPD exacerbation at Stavanger University Hospital, or at Dalane Medical Center (DMC) in Egersund, or who had tele-monitoring at home under outpatient treatment for acute COPD deterioration during a pilot project period (16th April 2010 - 31st December 2011)
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Frequency of hospital re-admissions due to COPD exacerbations during 12 months follow-up after TVC, as compared to admissions due to COPD exacerbations during 12 months pre-TVC | 12 months from inclusion period 16th April 2010 to 31st December 2011
  Number of re-admissions in hospital due to COPD exacerbations during 12 months follow-up after TVC, as compared to number of hospital admissions caused by COPD exacerbations the 12 months preceding TVC

SECONDARY OUTCOMES:
Length of hospital stays (days in hospital) when re-admitted during 12 months follow-up after TVC, as compered to length of hospital stays due to COPD the year preceding TVC | 12 months after inclusion period from 16th April 2010 to 31st December 2011

OTHER OUTCOMES:
self-perception of safety (n, %) | 4 weeks after TVC at inclusion, inclusion period from 16th April 2010 to 31st December 2011
  Patient's self-perception of safety when discharged from hospital without TVC, as compared to discharged to TVC at home
Time to first re-admission for COPD exacerbation | Days to re-admission from end of TVC, 14 days after included during inclusion period from 16th April 2010 to 31st December 2011
  Days to first re-admission for COPD exacerbation during 12 months follow-up after TVC, as compared to days from last discharge from hospital during the last 12 months preceding TVC to the index stay followed by TVC

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Grundt, MD PhD, Study Chair — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway